CLINICAL TRIAL: NCT05325151
Title: A Randomized Controlled Trial Comparing a Genetic Counseling Patient Preference Intervention vs. Conventional Genetic Counseling for Women at Elevated Risk for Breast Cancer
Brief Title: Genetic Counseling Patient Preference Intervention Versus Conventional Genetic Counseling for Women at Elevated Risk for Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Sweet, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-22013; NCI-2022-01136 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA248739 (NIH)
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Genetic Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (GCPP intervention) (Experimental): Patients receive GCPP intervention consisting of a series of educational videos on pre-genetic test information.
  Interventions: Other: Educational Intervention; Other: Survey Administration
- Arm II (conventional genetic counseling) (Active Comparator): Patients receive conventional genetic counseling.
  Interventions: Other: Genetic Counseling; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive GCPP intervention videos
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (GCPP intervention)
Other: Genetic Counseling — Receive genetic counseling
  Arms: Arm II (conventional genetic counseling)
Other: Survey Administration — Ancillary studies

SUMMARY:
This stage I clinical trial compares a genetic counseling patient preference (GCPP) intervention via EHR MyChart patient portal to conventional genetic counseling for women at elevated risk for breast cancer. Women at elevated breast cancer risk may be offered genetic counseling and genetic testing to further define whether they are at high risk (e.g. hereditary risk; BRCA mutation positive); moderate risk (e.g. risk based largely on family history and/or polygenic risk score) or average risk (e.g. general population). Genetic counseling may improve basic genetic knowledge, produce more accurate risk perceptions and tailor recommendations for greater perceived personal control regarding breast cancer risk. A single approach to genetic counseling may not fit the needs for all patients, and genetic counseling models that increase access to genetic testing and are more patient-centered may better serve patients. This trial may help researchers determine if a GCPP intervention can take the place of conventional genetic counseling, while being non-inferior in terms of adherence to screening recommendations, breast cancer genetic knowledge, accurate perception of risk, breast cancer-specific worry, and satisfaction with counseling compared to conventional genetic counseling. Study results will provide the efficacy for using a novel cancer genetic counseling approach via EHR MyChart patient portal that will be readily adaptable to other health care systems in the future, inform best practices, and reduce workforce burden.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the efficacy of genetic counseling patient preference (GCPP) compared to conventional genetic counseling for adherence to National Comprehensive Cancer Network (NCCN) guidelines for having: 1) a clinical encounter every 6-12 months; and 2) an annual mammogram (and breast magnetic resonance imaging [MRI] with contrast if recommended).

II. Determine the efficacy of the GCPP compared to conventional genetic counseling for adherence to other NCCN recommended cancer screening (e.g. colorectal cancer screening).

III. Determine the efficacy of the GCPP compared to conventional genetic counseling on breast cancer genetic knowledge, the accurate perception of breast cancer risk, breast cancer-specific worry, post-test/counseling distress, and satisfaction with counseling.

EXPLORATORY OBJECTIVE:

I. Explore the genetic counseling preferences among the GCPP group.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive GCPP intervention which uses REDCap and the MyChart patient portal to: 1) deliver a series of educational videos on pre-genetic test information; 2) provide multigene and polygenic risk score (PRS) test results; 3) obtain information about patients' questions/concerns about test results to use in post-genetic test counseling; and 4) determine patient preference (e.g. telehealth) for receipt of post-genetic test counseling.

ARM II: Patients receive conventional genetic counseling with utilization of multigene and polygenic risk score (PRS) test results.

ELIGIBILITY:
Inclusion Criteria:

* Being female.
* Ages 30-64.
* Being an Ohio State University (OSU) patient who uses MyChart.
* Undergoing routine screening mammography.
* Normal BI-RADS1.
* At elevated breast cancer risk by the Cancer Risk Assessment (CRA) tool.
* Able to read and speak English.
* Provide consent.

Exclusion Criteria:

* Previous genetic counseling.
* Previous genetic testing for cancer risk or known mutation in a breast cancer gene: ATM, BARD1, BRCA1, BRCA2, CDH1, CHEK2, NBN, PALB2, PTEN, TP53.
* Previous diagnosis of breast or ovarian cancer or personal history of lobular carcinoma in situ (LCIS) or breast hyperplasia (with or without atypia).
* Being a member of a focus group that assisted with the development of the intervention.

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 874 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to National Comprehensive Cancer Network (NCCN) guidelines of having a clinical encounter every 6-12 months | Up to 14 months
  Non-inferiority will be assessed by constructing a one-sided 95% confidence interval for the effect of genetic counseling patient preference (GCCP) versus conventional counseling and comparing the bound to a non-inferiority margin. Will use mixed effects logistic regression with adherence as the outcome, random intercept effects for genetic counselors, and fixed effects for study arm, breast cancer knowledge, breast cancer worry, post-test/counseling distress, and perception of breast cancer risk.
Adherence to NCCN guidelines of having an annual mammogram (and breast magnetic resonance imaging [MRI] with contrast if recommended) | Up to 14 months
  Non-inferiority will be assessed by constructing a one-sided 95% confidence interval for the effect of GCCP versus conventional counseling and comparing the bound to a non-inferiority margin. Will use mixed effects logistic regression with adherence as the outcome, random intercept effects for genetic counselors, and fixed effects for study arm, breast cancer knowledge, breast cancer worry, post-test/counseling distress, and perception of breast cancer risk.
Risk perception | Up to 14 months
  Determine the efficacy of the GCPP compared to conventional genetic counseling on breast cancer genetic knowledge, the accurate perception of breast cancer risk, breast cancer-specific worry, post-test/counseling distress, and satisfaction with counseling. Non-inferiority will be assessed by constructing a one-sided 95% confidence interval for the effect of GCCP versus conventional counseling and comparing the bound to a non-inferiority margin.
Breast cancer-specific worry | Up to 14 months
  Determine the efficacy of the GCPP compared to conventional genetic counseling on breast cancer genetic knowledge, the accurate perception of breast cancer risk, breast cancer-specific worry, post-test/counseling distress, and satisfaction with counseling. Non-inferiority will be assessed by constructing a one-sided 95% confidence interval for the effect of GCCP versus conventional counseling and comparing the bound to a non-inferiority margin.
Post-test/counseling distress | Up to 14 months
  Determine the efficacy of the GCPP compared to conventional genetic counseling on breast cancer genetic knowledge, the accurate perception of breast cancer risk, breast cancer-specific worry, post-test/counseling distress, and satisfaction with counseling. Non-inferiority will be assessed by constructing a one-sided 95% confidence interval for the effect of GCCP versus conventional counseling and comparing the bound to a non-inferiority margin.
Satisfaction with counseling | Up to 14 months
  Determine the efficacy of the GCPP compared to conventional genetic counseling on breast cancer genetic knowledge, the accurate perception of breast cancer risk, breast cancer-specific worry, post-test/counseling distress, and satisfaction with counseling. Non-inferiority will be assessed by constructing a one-sided 95% confidence interval for the effect of GCCP versus conventional counseling and comparing the bound to a non-inferiority margin.

SECONDARY OUTCOMES:
Adherence to other National Comprehensive Cancer Network (NCCN) recommended cancer screening (e.g. colorectal cancer screening) | Up to 14 months
  Non-inferiority will be assessed by constructing a one-sided 95% confidence interval for the effect of GCCP versus conventional counseling and comparing the bound to a non-inferiority margin.

OTHER OUTCOMES:
Genetic counseling preferences | Up to 14 months
  Will estimate the proportion of subjects who choose the remote (versus in-person) mode of the GCCP stratified by detection of high-risk variants, and construct 95% two-sided confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Sweet, MS, LGC, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sweet K, Reiter PL, Schnell PM, Senter L, Shane-Carson KP, Aeilts A, Cooper J, Spears C, Brown J, Toland AE, Agnese DM, Katz ML. Genetic counseling and testing for females at elevated risk for breast cancer: Protocol for the randomized controlled trial of the Know Your Risk intervention. Contemp Clin Trials. 2023 Oct;133:107323. doi: 10.1016/j.cct.2023.107323. Epub 2023 Sep 1. PMID 37661005
- See also: The Jamesline — http://cancer.osu.edu